CLINICAL TRIAL: NCT06840873
Title: Effectiveness of a 8-week Tele-Rehabilitative Exercise Training Program on Fatigue, Symptom Severity, and Quality of Life in Nurses With Long COVID: A Randomized Controlled Trial
Brief Title: Tele-Rehabilitative Exercise Training Program in Nurses With Long COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shang-Lin Chiang (Other)
Responsible Party: Sponsor-Investigator, Shang-Lin Chiang, Attending physician, National Defense Medical Center, Taiwan
Organization: National Defense Medical Center, Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: c202305117
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-01

CONDITIONS: Cardiorespiratory Fitness; Exercise; Long COVID; Nurses; Quality of Life (QOL); Fatigue; Stress; Tele-rehabilitation
MeSH Terms: conditions — Motor Activity; Post-Acute COVID-19 Syndrome; Fatigue | interventions — Wearable Electronic Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health consultation (Placebo Comparator): The participants with healthy consultation do aerobic training at home
  Interventions: Behavioral: Healthy consulation
- wearable device (Experimental): The participants with wearable device do exercise training at home
  Interventions: Device: wearable device

INTERVENTIONS:
Device: wearable device — Participants wore a knee brace with a sensor module on one side of the leg, the sensor could connect with the KNEESUP care APP which were installed in participant's mobile phone. The APP was designed with an individualized exercise program and the knee brace sensor could detect the action moment of the participants during exercise. This equipment could help the participants to achieve professional-level home rehabilitation, including 3 aerobic and 2 strengthening exercise sessions per week at a moderate intensity, 30 min/session.
  Arms: wearable device
Behavioral: Healthy consulation — Participants received routine outpatient health education.
  Arms: Health consultation

SUMMARY:
Long COVID can cause a decline in cardiorespiratory fitness, resulting in fatigue and negative impacts on individuals' quality of life (QoL), particularly in nurses who play a crucial role in public health. Combining with reduced cardiorespiratory fitness and suffering from a spectrum of long-COVID symptoms might substantially exaggertate fatigue, perceived stress, and reduce willingness to work for hospital nurses. Therefore, this study aimed to evaluate the effectiveness of tele-rehabilitative exercise on fatigue, perceived stress, symptom severity of long COVID, and QoL in this population.

DETAILED DESCRIPTION:
The intervention is an extra 8-week tele-rehabilitative exercise program (3 aerobic and 2 strengthing exercise sessions/week at a moderate intensity, 30 min/session), monitored through a wearable devices and a mobile App. The evaluation of the rehabilitation results can be presented as a data chart, and the treatment effects are also clearly presented. Outcome measures were assessed at baseline, 4, and 8 weeks. Cardiorespiratory fitness was measured before and after the intervention via cardiopulmonary exercise tests.

ELIGIBILITY:
Inclusion Criteria:

* nurses older than 20 years of age
* have reported a positive result on a COVID-19 rapid test or nucleic acid test
* one or more of the following symptoms for more than four weeks: fatigue, discomfort after physical or mental exertion, fever, cardiopulmonary symptoms such as difficulty breathing or shortness of breath, cough, chest pain, or palpitations (CDC, 2022)
* able to perform activities independently without assistance
* total score of 36 or higher on the Fatigue Severity Scale (FSS), confirming fatigue symptoms, and report that these symptoms either appeared after the infection or worsened following the infection

Exclusion Criteria:

* without the equipment to install a mobile application (APP)
* unsuitable for wearing devices due to any leg diseases
* unable to engage in aerobic or strength training due to neurological or musculoskeletal disorders
* pregnancy
* cancer
* absolute and relative contraindications for cardiopulmonary testing or exercise training
* unsuitable for participation in this study by a rehabilitation specialist;
* regular exercisers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Fatigue (score) | 10 minutes
  The Chinese version of the Fatigue Severity Scale (CFSS) (Wang et al., 2016) assesses the severity of fatigue in the participants. The scale is a self-administered questionnaire. The scale evaluates the severity of fatigue symptoms and their impact on daily activities over the past two weeks. It consists of 9 items, rated on a 7-point scale, with scores ranging from 1 to 7, where 1 indicates strong disagreement and 7 indicates strong agreement. The minimum score is 9, and the maximum score is 63. Higher scores indicate more severe fatigue, with a total score of 36 (inclusive) or higher indicating severe fatigue.
O2 pulse in ml/beat | 30 minutes
  It means the heart pumps O2 volume by each heart beat, and also means left ventricle function.
Aerobic capacity (VO2 max in ml/kg/min ) | 30 minutes
  Maximal VO2 during testing, also means aerobic capacity
Working load in watt | 30 minutes
  Maximal Working load during testing
Heart rate recovery in beat/min | 30 minutes
  Heart rate recovery is measured by recording your heart rate immediately after stopping exercise, and then at intervals (e.g., 1 minute and 2 minutes) after the exercise ends, which reflects autonomic nervous system function.
Anaerobic threshold (AT in ml/kg/min) | 30 minutes
  The point during exercise at which lactate (a byproduct of anaerobic metabolism) starts to accumulate in the blood faster than it can be removed. This indicates a shift from primarily aerobic energy production to more anaerobic energy production.
Severity of long COVID symptoms (scores) | 10 minutes
  This study uses the Chinese version of the Post-COVID-19 Functional Status Scale (PCFS) translated by Liao and Cheng (2023), which was originally developed by Frederikus A. Klok. It assesses changes in daily living, work and study activities, social activities, and overall functional status over the past week (Klok et al., 2020). The scale consists of two parts: the functional status scale and the symptom checklist. The first part, the functional status scale, is divided into five levels from 0 to 4. The second part, the post-infection symptom checklist, checks for specific symptoms that appear after COVID-19 infection. It is divided into five levels. This checklist evaluates respiratory, cardiovascular, gastrointestinal, neurological, psychological, and musculoskeletal symptoms.

SECONDARY OUTCOMES:
Quality of life (scores) | baseline, 4, and 8 weeks
  The indicator of quality of life in this study will use Taiwan Concise Version of the World Health Organization Quality of Life Questionnaire (WHOQOL) to evaluate. The Taiwan version development team led by Yao Kaiping developed a brief version of the questionnaire (WHOQOL-BREF) based on WHOQOL-100. The questionnaire includes 1 question measuring the overall quality of life, 1 question measuring general health, and 7 questions measuring the physical domain. , 6 questions measure the psychological domain (psychological domain), 3 questions measure the social relationship domain (social relationships domain), and 8 questions measure the environment domain (environment domain), and add 1 local question to the social relationship and environment domains, totaling 28 questions. The item is a 5-point scale, with higher scores indicating a higher quality of life. The total score ranges from 25 to 140.
Perceived stress (scores) | baseline, 4, and 8 weeks
  The Chinese version of the Perceived Stress Scale (PSS) measures the perception of stress (Chiu, 2012). The original scale was developed by Cohen et al. (Cohen et al., 1983). The Chinese version has shown good reliability and validity in a study of nurses in Taiwan, with a Cronbach's alpha of 0.73. The scale is a self-administered questionnaire that measures the level of perceived stress in the past month. It consists of 14 items, all rated using a Likert scale with five response options: "Never," "Occasionally," "Sometimes," "Often," and "Always" (0-4 points). Seven of the items (4, 5, 6, 7, 9, 10, 13) are positive questions that need to be reverse-scored. The total score ranges from 0 to 56, with higher scores indicating higher perceived stress. A score of 0-28 is considered within the normal stress range, 29-37 indicates high stress, and 38-56 suggests the need to seek external support.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-service General Hospital, Tiapei, Taiwan

IPD SHARING:
Plan to Share IPD: No